CLINICAL TRIAL: NCT04108676
Title: a Single-center, One-arm, Open, and Fixed Sequences Study to Evaluate the Effects of Omeprazole on the Pharmacokinetics of Fluzoparib in Healthy Male Volunteers
Brief Title: Effect of Omeprazole on PK of Fluzoparib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FZPL-I-111
Record Dates: First submitted 2019-09-19; First posted 2019-09-30 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2021-09

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — fluzoparib; Omeprazole

STUDY DESIGN:
Intervention Model Description: repeated oral doses of Omeprazole on the pharmacokinetic profile of a single dose of Fluzoparib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Drug: Fluzoparib Drug: Omeprazole
  Interventions: Drug: Fluzoparib; Drug: Omeprazole

INTERVENTIONS:
Drug: Fluzoparib — PARP inhibitor
Drug: Omeprazole — proton pump inhibitor

SUMMARY:
The purpose of this study is to evaluate the Effect of Omeprazole on the Pharmacokinetics of Fluzoparib in Healthy male Adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years (including both ends), male;
2. Male volunteers have a body weight ≥ 50.0 kg and a body mass index (BMI) between 19 and 28 kg/m2 (including both ends);
3. Male volunteers are willing to have no birth plans in the next 6 months and voluntarily take effective contraceptive measures;
4. Volunteers voluntarily sign written informed consent.

Exclusion Criteria:

1. Previous or currently suffering from circulatory system (myocarditis, coronary heart disease, pathological arrhythmia, stroke, etc.), endocrine system, nervous system, digestive system (peptic ulcer, colitis, pancreatitis, etc.), respiratory system (Invasive lung disease, pneumonia, dyspnea, etc., urogenital system (chronic kidney disease, renal insufficiency, renal anemia), hematology, immunology, psychiatry and metabolic abnormalities, etc. Result of any other disease;
2. A history of allergies to drugs, foods or other substances; allergies, including a history of severe drug allergies or drug allergies; a history of allergies to Fluzoparib capsules or omeprazole magnesium enteric-coated tablets
3. Those who have undergone surgery within 4 weeks prior to the trial or who plan to undergo surgery during the study;
4. Those who have taken any drugs or health care products (including Chinese herbal medicines) within 14 days before the test;
5. Any drug that inhibits or induces liver metabolism of the drug within 30 days prior to the test (eg, inducer - barbiturate, carbamazepine, phenytoin, glucocorticoid, omeprazole; inhibitor - SSRI resistance) Depressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines;
6. Those who participated in any clinical trial and took any clinical trial drug within 3 months prior to the trial;
7. Donate blood or massive blood loss (≥200 mL), receive blood transfusion or use blood products within 3 months before enrollment;
8. One or more non-pharmaceutical contraceptives cannot be used during the volunteer trial;
9. Those who have special requirements for diet and cannot follow the unified diet;
10. Drink excessive amounts of tea, coffee and/or caffeinated beverages (8 cups or more, 1 cup = 250 mL) per day;
11. smokers or smokers with more than 5 cigarettes per day for the first 3 months of the trial or who cannot stop using any tobacco products during the trial period;
12. Alcoholics or those who regularly drink alcohol within 6 months prior to the test, ie drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) or during the test period Stop using any alcoholic products;
13. Drug abusers or soft drugs (eg marijuana) 3 months prior to the trial or hard drugs (eg cocaine, phencyclidine, etc.) 1 year prior to the trial; and nicotinic positive volunteers
14. Abnormal vital signs (systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure <50 mmHg or >90 mmHg; pulse <50 bpm or >100 bpm) or physical examination, electrocardiogram, laboratory examination, imaging examination abnormalities Clinically significant (subject to the judgment of the clinical research doctor);
15. have a history of dysphagia or any history of gastrointestinal disease that affects drug absorption;
16. Those who have undergone any surgery within the first 6 months of screening; have previously undergone any surgery that affects gastrointestinal absorption (including gastrectomy, bowel resection, stomach reduction surgery, etc.);
17. The volunteer refused to discontinue any beverage containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or any juice, 48 hours before the study drug was administered until the end of the study;
18. Creatinine clearance (CLCr) <80 mL/min, or creatinine above the upper limit of normal;
19. Volunteers may not be able to complete the study for other reasons or those the investigator believes should not be included.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Fluzoparib: | through study completion, up to 24 weeks
  Cmax
Area Under the Plasma Concentration-Time Curve From 0 to t of Fluzoparib: | through study completion, up to 24 weeks
  AUC0-t
Area Under the Plasma Concentration-Time Curve From 0 to infinity of Fluzoparib: | through study completion, up to 24 weeks
  AUC0-∞ (if available)

SECONDARY OUTCOMES:
Safety in terms of Adverse Events Assessments | through study completion, up to 24 weeks
  Adverse Events Assessments (NCI-CTC AE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, PhD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The third xiangya hospital Hospital,of central south university, Changsha, Hunan, China

REFERENCES:
- [Derived] Li L, Xiang YX, Yang GP, Zhang XF, Yang XY, Yang S, Huang J. Pharmacokinetic effects of proton pump inhibitors on the novel PARP inhibitor fluzoparib: a single-arm, fixed-sequence trial in male healthy volunteers. Invest New Drugs. 2021 Jun;39(3):796-802. doi: 10.1007/s10637-020-01034-w. Epub 2021 Jan 9. PMID 33420642